CLINICAL TRIAL: NCT03866538
Title: Open-label Withdrawal Trial of Budesonide in Patients With Immune Mediated Enteropathies
Brief Title: Budesonide in Patients With Immune Mediated Enteropathies
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study recruitment was difficult and not acheived
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joseph A. Murray, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-008639
Record Dates: First submitted 2019-02-27; First posted 2019-03-07 (Actual); Results first posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Enteropathy; Celiac Disease; CVID Enteropathy; Collagenous Sprue; Autoimmune Enteropathy
MeSH Terms: conditions — Intestinal Diseases; Celiac Disease; Collagenous Sprue; Autoimmune enteropathy

STUDY DESIGN:
Intervention Model Description: Randomized, open-label withdrawal of budesonide versus continued budesonide therapy in patients with immune-mediated enteropathies that have had symptomatic and histologic improvement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Continued Budesonide (No Intervention): Patients in this arm continue budesonide at the dose they were taking at the time of enrollment in the trial
- Withdrawal of Budesonide (Experimental): Patients are weaned off of budesonide over 2 weeks and continued off of the medication for the duration of the trial
  Interventions: Drug: Withdrawal of Oral Budesonide

INTERVENTIONS:
Drug: Withdrawal of Oral Budesonide — The intervention arm will taper and stop budesonide therapy (withdrawal).
  Arms: Withdrawal of Budesonide

SUMMARY:
Researchers are trying to determine if withdrawal of budesonide therapy in patients with immune-mediated enteropathies doing well on therapy will result in worsening symptoms, histology, quality of life, and micronutrient/nutritional status when compared to continued therapy.

DETAILED DESCRIPTION:
This study aims to evaluate patients with small intestinal diseases caused by the immune system (refractory celiac disease type 1, CVID enteropathy, autoimmune enteropathy, and collagenous enteropathy) who have had improvement in symptoms and small intestine healing with oral budesonide.

Patients who meet inclusion criteria and agree to enter the study will be included for 12 weeks or until they choose to discontinue or there are concerns for safety.

At the beginning of the study, patients will undergo questionnaires, blood draw, urine and stool collections, physical exam, and an upper scope (esophagogastroduodenoscopy) with biopsies from the small intestine. They will then be randomized to either continued therapy on their current dose and formulation of budesonide (medication provided by the study) or to withdrawal of the medication over 2 weeks and then no medication during the study. Daily questionnaire on symptoms will be recorded.

Patients will be assessed in the clinical research unit monthly during the study with a questionnaire, physical exam, blood draw, and urine/stool collections.

Finally, at the end of the trial (12 weeks) or at the time of withdrawal from the trial, the patients will complete questionnaires, physical exam, blood collection, urine/stool collection, and upper scope (esophagogastroduodenoscopy) with small bowel biopsies.

ELIGIBILITY:
Inclusion Criteria

* Patients will be recruited from the Division of Gastroenterology and Hepatology and the Mayo Clinic in Rochester, MN.
* Adult patients with immune mediated enteropathies who have had improvement in symptoms and histology on oral budesonide therapy.

Exclusion Criteria

* Age <18 years
* Positive stool gluten testing in patients with refractory celiac disease
* Small bowel malignancy or history of small bowel malignancy
* Refractory celiac disease type 2
* Post-transplant lymphoproliferative disorder associated enteropathy
* No prior improvement in symptoms and histology with budesonide therapy
* Discontinuation of budesonide therapy prior to the trial
* Other concurrent systemic corticosteroids
* Other immune mediating medications, for example but not limited to azathioprine, 6-mercaptopurine, cyclosporine, methotrexate, anti-TNF monoclonal antibodies, alpha-4 beta-7 integrin inhibiting monoclonal antibody, interleukin 12/23 inhibiting monoclonal antibody, JAK inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Murray, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ludvigsson JF, Leffler DA, Bai JC, Biagi F, Fasano A, Green PH, Hadjivassiliou M, Kaukinen K, Kelly CP, Leonard JN, Lundin KE, Murray JA, Sanders DS, Walker MM, Zingone F, Ciacci C. The Oslo definitions for coeliac disease and related terms. Gut. 2013 Jan;62(1):43-52. doi: 10.1136/gutjnl-2011-301346. Epub 2012 Feb 16. PMID 22345659
- [Background] Choung RS, Unalp-Arida A, Ruhl CE, Brantner TL, Everhart JE, Murray JA. Less Hidden Celiac Disease But Increased Gluten Avoidance Without a Diagnosis in the United States: Findings From the National Health and Nutrition Examination Surveys From 2009 to 2014. Mayo Clin Proc. 2016 Dec 5:S0025-6196(16)30634-6. doi: 10.1016/j.mayocp.2016.10.012. Online ahead of print. PMID 28017411
- [Background] Leffler DA, Dennis M, Hyett B, Kelly E, Schuppan D, Kelly CP. Etiologies and predictors of diagnosis in nonresponsive celiac disease. Clin Gastroenterol Hepatol. 2007 Apr;5(4):445-50. doi: 10.1016/j.cgh.2006.12.006. Epub 2007 Mar 26. PMID 17382600
- [Background] Rubio-Tapia A, Murray JA. Classification and management of refractory coeliac disease. Gut. 2010 Apr;59(4):547-57. doi: 10.1136/gut.2009.195131. PMID 20332526
- [Background] Mukewar SS, Sharma A, Rubio-Tapia A, Wu TT, Jabri B, Murray JA. Open-Capsule Budesonide for Refractory Celiac Disease. Am J Gastroenterol. 2017 Jun;112(6):959-967. doi: 10.1038/ajg.2017.71. Epub 2017 Mar 21. PMID 28323276
- [Background] Greenberg GR, Feagan BG, Martin F, Sutherland LR, Thomson AB, Williams CN, Nilsson LG, Persson T. Oral budesonide for active Crohn's disease. Canadian Inflammatory Bowel Disease Study Group. N Engl J Med. 1994 Sep 29;331(13):836-41. doi: 10.1056/NEJM199409293311303. PMID 8078529
- [Background] Campieri M, Ferguson A, Doe W, Persson T, Nilsson LG. Oral budesonide is as effective as oral prednisolone in active Crohn's disease. The Global Budesonide Study Group. Gut. 1997 Aug;41(2):209-14. doi: 10.1136/gut.41.2.209. PMID 9301500
- [Background] Tremaine WJ, Hanauer SB, Katz S, Winston BD, Levine JG, Persson T, Persson A; Budesonide CIR United States Study Group. Budesonide CIR capsules (once or twice daily divided-dose) in active Crohn's disease: a randomized placebo-controlled study in the United States. Am J Gastroenterol. 2002 Jul;97(7):1748-54. doi: 10.1111/j.1572-0241.2002.05835.x. PMID 12135030
- [Background] Rubio-Tapia A, Malamut G, Verbeek WH, van Wanrooij RL, Leffler DA, Niveloni SI, Arguelles-Grande C, Lahr BD, Zinsmeister AR, Murray JA, Kelly CP, Bai JC, Green PH, Daum S, Mulder CJ, Cellier C. Creation of a model to predict survival in patients with refractory coeliac disease using a multinational registry. Aliment Pharmacol Ther. 2016 Oct;44(7):704-14. doi: 10.1111/apt.13755. Epub 2016 Aug 3. PMID 27485029
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Continued Budesonide: Patients in this arm continued budesonide at the dose they were taking at the time of enrollment in the trial
- Withdrawal of Budesonide: Patients were weaned off of budesonide over 2 weeks and continued off of the medication for the duration of the trial
  Withdrawal of Oral Budesonide: The intervention arm tapered and stoped budesonide therapy (withdrawal).
Period: Overall Study
Arm/Group | Continued Budesonide | Withdrawal of Budesonide
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated due to recruitment being difficult and not achieved
Groups:
- Total: Total of all reporting groups
Arm/Group | Continued Budesonide | Withdrawal of Budesonide | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 1 | 1
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Histology
Description: Investigators will determine change in small bowel villi after withdrawal of budesonide compared to continued therapy to assess small intestinal injury. This will be accomplished by esophagogastroduodenoscopy (upper scope) with biopsies from the small intestine.
Time Frame: 12 weeks
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Continued Budesonide | Withdrawal of Budesonide
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Symptoms
Description: Symptoms (monitored daily) will be compared between patients that withdraw from budesonide compared to those that continue budesonide therapy. Symptoms will be measured on the Celiac Disease Symptom Diary (CDSD) questionnaire. First question asks if subject has diarrhea and how many times. Second question asks if subject has spontaneous bowel movement and how many. Third question asks if subject had abdominal pain and to rate on a scale from 0 to 10 with higher numbers being worse pain. Fourth question asks if experiencing bloating and if it is very mild, mild, moderate, severe, or very severe. Fifth question asks if subject has nausea and if it is ranked very mild, mild, moderate, severe, or very severe. The sixth question asks if the subject has experienced tiredness and to rank very mild, mild, moderate, severe or very severe. Each question is evaluated for changes or trends over time, and a composite score including multiple questions can be calculated and compared.
Time Frame: 12 weeks
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Continued Budesonide | Withdrawal of Budesonide
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Quality of Life: Celiac Disease Quality of Life Questionnaire (CD-QOL)
Description: Quality of life will be assessed monthly comparing those that withdraw from budesonide compared to those that continue therapy. This will be assessed by the Celiac Disease Quality of Life Questionnaire (CD-QOL). This survey includes 20 questions with scores for each ranging from 1 to 5, with higher numbers indicating improved quality of life. Total scores will range from 20 to 100 with higher numbers indicating better quality of life.
Time Frame: 12 weeks
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Continued Budesonide | Withdrawal of Budesonide
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Weight
Description: Weight in kilograms will be monitored throughout the study. Changes will be compare between those withdrawing from budesonide compared to those continuing therapy.
Time Frame: 12 weeks
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Continued Budesonide | Withdrawal of Budesonide
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Iron
Description: Iron in the blood will be compared to those that withdraw from budesonide compared to those that continue therapy. This will be assessed at the initiation and completion of the trial.
Time Frame: 12 weeks
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Continued Budesonide | Withdrawal of Budesonide
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Vitamin D
Description: 25-hydroxy vitamin D in the blood will be compared to those that withdraw from budesonide compared to those that continue therapy. This will be assessed at the initiation and completion of the trial.
Time Frame: 12 weeks
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Continued Budesonide | Withdrawal of Budesonide
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Vitamin B12
Description: Vitamin B12 in the blood will be compared to those that withdraw from budesonide compared to those that continue therapy. This will be assessed at the initiation and completion of the trial.
Time Frame: 12 weeks
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Continued Budesonide | Withdrawal of Budesonide
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Folate
Description: Folate in the blood will be compared to those that withdraw from budesonide compared to those that continue therapy. This will be assessed at the initiation and completion of the trial.
Time Frame: 12 weeks
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Continued Budesonide | Withdrawal of Budesonide
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Zinc
Description: Zinc in the blood will be compared to those that withdraw from budesonide compared to those that continue therapy. This will be assessed at the initiation and completion of the trial.
Time Frame: 12 weeks
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Continued Budesonide | Withdrawal of Budesonide
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in Copper
Description: Copper in the blood will be compared to those that withdraw from budesonide compared to those that continue therapy. This will be assessed at the initiation and completion of the trial.
Time Frame: 12 weeks
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Continued Budesonide | Withdrawal of Budesonide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 2 weeks
Description: Study was terminated due to recruitment being difficult and not achieved. There was no accrual in the Continued Budesonide arm
Arm/Group | Continued Budesonide | Withdrawal of Budesonide
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continued Budesonide (N=0) | Withdrawal of Budesonide (N=1)
Diarrhea (Gastrointestinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study was terminated due to recruitment being difficult and not achieved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT03866538/Prot_SAP_000.pdf